CLINICAL TRIAL: NCT01165463
Title: RCT of Two Speed of Processing Modes to Prevent Cognitive Decline in Older Adults
Brief Title: Iowa Healthy and Active Minds Study
Acronym: IHAMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fredric D Wolinsky (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor-Investigator, Fredric D Wolinsky, Professor of Public Health, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 200908789; 1RC1AG035546-01 (NIH)
Record Dates: First submitted 2010-07-13; First posted 2010-07-19 (Estimated); Last update posted 2019-06-21 (Actual); Status verified 2019-06

CONDITIONS: Visual Processing Speed
Keywords: Aging; Healthy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Clinic-based SOPT basic training (Experimental): Clinic-based SOPT basic training for 10 hours.
  Interventions: Behavioral: SOPT basic training
- Home-based SOPT basic training (Experimental): Home-based SOPT basic training for 10 hours.
  Interventions: Behavioral: SOPT basic training
- Crossword Puzzles Training (Active Comparator): Crossword puzzles training for 10 hours in our lab.
  Interventions: Behavioral: Crossword Puzzles
- SOPT basic and SOPT booster-training (Experimental): Clinic-based SOPT basic training and SOPT booster training.
  Interventions: Behavioral: SOPT basic training; Behavioral: SOPT booster training

INTERVENTIONS:
Behavioral: SOPT basic training — 10 hours of basic training
  Arms: Clinic-based SOPT basic training; Home-based SOPT basic training; SOPT basic and SOPT booster-training
Behavioral: Crossword Puzzles — Subjects train with puzzles 10 hrs in lab.
  Arms: Crossword Puzzles Training
Behavioral: SOPT booster training — 4 hours of subsequent booster-training
  Arms: SOPT basic and SOPT booster-training

SUMMARY:
This is second-generation study based on results from ACTIVE (Advanced Cognitive Training for Independent and Vital Elderly). This four-arm study is known as IHAMS (the Iowa Healthy and Active Minds Study). The investigators will formally test from an intent-to-treat perspective for differences on the primary and secondary outcomes based on whether participants were randomized to the basic on-site speed of processing training (SOPT) group (G1), to the on-site basic SOPT plus subsequent booster-training group (G2), to the basic at-home SOPT group (G3), or to the basic attention-control group (G4). Basic training involves 10 hours of either the SOPT or attention-control training during the first 6 weeks of participation. Booster-training involves 4 additional hours of SOPT training at 11 months of participation.

DETAILED DESCRIPTION:
In this study, our specific aims are to conduct a randomized controlled trial (RCT) with one-year follow-up that can be fully completed within the NIH Challenge Grant two-year period. The goal of the RCT is to improve cognitive performance among older adults to enhance their quality of life now and into the future. We will randomize 600 participants to four treatment arms separately within two age strata (50-64, and 65 and older).

The four groups include: G1, basic on-site SOPT; G2, on-site basic SOPT plus subsequent booster-training group; G3, basic at-home SOPT; or G4, basic attention-control group. Basic training involves 10 hours of either the SOPT or attention-control training during the first 6 weeks of participation. Booster-training involves 4 additional hours of SOPT training at 11 months of participation.

Our primary outcome measure is speed of processing, and we will use several reliable and valid instruments to provide a multidimensional assessment, including the Useful Field of View Test, the Symbol Digit Modalities Test, the Trail Making Test, the Controlled Oral Word Association Test, the Digit Vigilance Test, and the Stroop Color and Word Test.

There are seven key hypotheses (Hn). H1 involves a replication of ACTIVE (i.e., on-site SOPT delivery, with or without booster-training) in which groups G1 and G2 are combined vs. the attention control group and hypothesizes statistically significant evidence to support the benefit of being assigned to on-site training vs. the attention control group.

H2 and H3 are designed to separate the basic training effect (H2) from the basic plus booster-training effect (H3) among the on-site delivery groups (G1 and G2) vs. the attention control group (G4), and hypothesizes benefits of SOPT training vs. attention control regardless of booster-training.

H4 represents the test of the at-home delivery of SOPT training (G3) vs. the attention control group (G4). H4 hypothesizes that there will be statistically significant evidence indicating the benefit of being assigned to G3 (at-home training) vs. the attention control group (G4).

H5 and H6 evaluate the different modes of implementing the speed of processing intervention. H5 represents a head-to-head comparison of the basic on-site delivery vs. the at-home delivery of the SOPT intervention. H5 hypothesizes that the effect of at-home SOPT training (G3) will be greater than the effect of on-site SOPT training (G1).

H6 represents a head-to-head comparison of the on-site basic plus booster SOPT training (G2) vs. the at-home delivery of the SOPT intervention. H6 hypothesizes that the effect for at-home SOPT (G3) will be larger than that for the on-site SOPT with booster-training group (G2).

Finally, H7 represents the head-to-head test of on-site basic SOPT (G1) to on-site basic plus booster training SOPT group (G2) . H7 hypothesizes that the difference between the two will reflect the value of booster training.

The investigators will replicate all of the above analyses within each age strata (50-64 vs. > 65) and compare effect sizes across strata.

ELIGIBILITY:
Inclusion Criteria:

* 50 years of age or older
* Patient of the FCC in Family Medicine or General Internal Medicine Clinic at UIHC
* No known memory problems

Exclusion Criteria:

* Significant vision impairments
* Lack of access to a computer or owns a MAC
* Lives more than 37 miles from the lab
* Traumatic Brain Injury or severe stroke

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 681 (Actual)
Dates: Start 2009-09; Primary Completion 2011-12 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Useful Field of View Test | 12 months
  The Useful Field of View (UFOV) is a computer-administered test of functional vision and visual attention. UFOV consists of three subtests which assess speed of visual processing under increasingly complex task demands. The examinee must detect, identify, and localize briefly presented targets.

SECONDARY OUTCOMES:
Digit Vigilance Test | 12 months
  Subject crosses out all 6's on an 8 x 11.5 page of random numbers while being timed.
Symbol Digit Modalities Test | 12 Months
  Subject matches a number to a symbol corresponding to a key on the top of the page. They are timed and allowed 90 to complete.
Controlled Oral Word Association Test | 12 Months
  Subject states all the ordinary words they can think of that start with the letter C while being timed for 60 seconds. They repeat this task with the letters F and L.
Comprehensive Trail Making Test | 12 Months
  Both parts of the Trail Making Test consist of 25 circles distributed over a sheet of paper. In Part A, the circles are numbered 1 - 25, and the patient should draw lines to connect the numbers in ascending order. In Part B, the circles include both numbers (1 - 13) and letters (A - L); as in Part A, the patient draws lines to connect the circles in an ascending pattern, but with the added task of alternating between the numbers and letters (i.e., 1-A-2-B-3-C, etc.) They are timed until completion.
Stroop | 12 months
  Subject must read aloud. Part A- Read the words on the page, Part B - Read the colors on the page, and Part C - Say the color of the ink the words are printed in. Each part is timed giving subject 45 seconds per part.

CONTACTS AND LOCATIONS:
Overall Officials: Fredric D Wolinksy, Ph.D., Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wolinsky FD, Vander Weg MW, Howren MB, Jones MP, Martin R, Luger TM, Duff K, Goerdt C, Wolfe S, Dotson MM. Protocol for a randomised controlled trial to improve cognitive functioning in older adults: the Iowa Healthy and Active Minds Study. BMJ Open. 2011 Jan 1;1(2):e000218. doi: 10.1136/bmjopen-2011-000218. PMID 22021885
- [Result] Wolinsky FD, Vander Weg MW, Howren MB, Jones MP, Martin R, Luger TM, Duff K, Dotson MM. Interim analyses from a randomised controlled trial to improve visual processing speed in older adults: the Iowa Healthy and Active Minds Study. BMJ Open. 2011 Nov 21;1(2):e000225. doi: 10.1136/bmjopen-2011-000225. Print 2011. PMID 22106377
- [Result] Wolinsky FD, Vander Weg MW, Howren MB, Jones MP, Dotson MM. A randomized controlled trial of cognitive training using a visual speed of processing intervention in middle aged and older adults. PLoS One. 2013 May 1;8(5):e61624. doi: 10.1371/journal.pone.0061624. Print 2013. PMID 23650501
- [Result] Wolinsky FD, Vander Weg MW, Howren MB, Jones MP, Dotson MM. The effect of cognitive speed of processing training on the development of additional IADL difficulties and the reduction of depressive symptoms: results from the IHAMS randomized controlled trial. J Aging Health. 2015 Mar;27(2):334-54. doi: 10.1177/0898264314550715. Epub 2014 Sep 19. PMID 25239928
- [Derived] Wolinsky FD, Vander Weg MW, Howren MB, Jones MP, Dotson MM. Effects of cognitive speed of processing training on a composite neuropsychological outcome: results at one-year from the IHAMS randomized controlled trial. Int Psychogeriatr. 2016 Feb;28(2):317-30. doi: 10.1017/S1041610215001428. Epub 2015 Sep 14. PMID 26364892